CLINICAL TRIAL: NCT03048097
Title: Optimizing Acquisition Parameters and Interpretive Methods of FDG-PET/CT With Rb-82 Myocardial Perfusion Imaging for Evaluation of Cardiac Sarcoidosis
Brief Title: Optimizing Acquisition Parameters and Interpretive Methods of FDG-PET/CT With Rb-82
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1512016912
Record Dates: First submitted 2017-02-02; First posted 2017-02-09 (Estimated); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis | interventions — Fluorodeoxyglucose F18; Rubidium

STUDY DESIGN:
Intervention Model Description: A comparison will be made between initial images, and images taken 2 weeks later of the same group of individuals.
Masking Description: images will be interpreted without identification
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- All Participants (Experimental): Subjects with high-likelihood of cardiac sarcoidosis.
  Interventions: Drug: Fluorodeoxyglucose; Drug: Rubidium; Diagnostic Test: FDG-PET/CT with Rb82 Myocardial Perfusion Imaging

INTERVENTIONS:
Drug: Fluorodeoxyglucose — a radiopharmaceutical used in the medical imaging modality positron emission tomography (PET)
  Other Names: FDG
Drug: Rubidium — used in PET scans
  Other Names: RB82
Diagnostic Test: FDG-PET/CT with Rb82 Myocardial Perfusion Imaging — A 18-20 gauge catheter equipped with a 3-way stopcock will be inserted preferably in the antecubital vein. Cardiac FDG-PET imaging will be performed on the YNHH GE Discovery ST PET/CT scanner following a high fat/low carbohydrate diet and a prolonged fast as is current clinical protocol. Resting ECG-gated dynamic Rb-82 PET imaging will be performed using 20-30 mCi of Rb82 as per YNHH clinical imaging protocol and established clinical guidelines. FDG-PET imaging will be performed following a high fat/low carbohydrate diet (instructions provided to patient) and a fast of greater than 12 hours. The patient will be injected with the same dose of FDG (8-10mCi) as they received for their index clinical examination. Cardiac FDG imaging will be performed using a single 3D acquisition over the heart. Low-dose CT images (120 kV, 50-150 mA based on BMI) for the purposes of attenuation correction will be performed before Rb82 and FDG imaging sequences.
  Other Names: FDG PET

SUMMARY:
In this this investigation, 15 subjects with a high probability of cardiac sarcoidosis based on clinical criteria and abnormal cardiac FDG uptake on initial, clinically indicted FDG PET study will be considered for this study. The study will test the following Aims:

Aim 1. Effect of FDG incubation time on visual and quantitative interpretation of FDG uptake.

Changes in incubation time can affect imaging target:background ratios and study sensitivity/specificity. For the study-directed exam, all patients will undergo sequential cardiacfocused FDG-PET imaging at 90 and 120 minutes after injection of FDG. Imaging variables will be evaluated as below.

Aim 2. Reproducibility of FDG and Rb82 PET findings on sequential imaging. It is unknown whether FDG-positive imaging findings in cardiac sarcoidosis are reproducible. All patients will undergo study-directed FDG-PET/CT with MPI imaging within approximately 2 weeks from initial clinical scan.

DETAILED DESCRIPTION:
Sarcoidosis is a systemic disease of unknown etiology characterized by non-caseating granulomatous inflammation. The pathophysiologic features of cardiac sarcoidosis include macrophage-induced, T-cell mediated non-caseating granulomatous inflammation, followed by myocardial scarring/fibrosis with clinical sequelae including arrhythmias, conduction abnormalities, and contractile dysfunction. These lead to high event rates in patients with cardiac sarcoidosis, with several studies reporting a prevalence of ventricular tachycardia ranging from 23% to 38% and an ~ 20% rate of clinical congestive heart failure.

FDG-PET/CT with Rb82 myocardial perfusion imaging (FDG-PET with MPI) is becoming the gold standard imaging technique for evaluating the degree of inflammation and the response to immunosuppressive treatment in patients with cardiac sarcoidosis. FDG PET imaging allows for evaluation of inflammatory macrophage infiltration, while Rb82 MPI allows for determination of myocardial scar burden. Despite emerging data from our center and others on the clinical utility of this technique in predicting prognosis, there is little consensus on the reproducibility of this technique or optimal imaging acquisition techniques and interpretative strategies.

In this study, patients with a high clinical likelihood of cardiac sarcoidosis will undergo a study-directed FDG PET/CT with Rb82 myocardial perfusion imaging study approximately 2 weeks following an initial clinically-directed examination.

The two FDG PET with MPI examinations will be examined for reproducibility of imaging findings, including: SUVmax, SUVmean, distribution of FDG uptake, extra cardiac FDG uptake, SUVvolume, SUVvolume:intensity, perfusion defect size/severity/location, LV ejection fraction, myocardial blood flow.

Strict attention will be paid to ensure patients undergo the same metabolic preparation prior to the two examinations.

ELIGIBILITY:
Inclusion Criteria:

Symptoms

* Palpitations/presyncope/syncope
* Heart failure symptoms Signs
* Abnormal ECG or Holter
* RBBB, LBBB, LAFB
* Abnormal Q waves in ≥2 leads
* 1st degree AVB > 240 msec, 2nd/3rd deg. AVB
* Frequent PVCs
* VT (sustained/non-sustained)
* LVEF < 50%
* Cardiac Regional Wall Motion Abnormality

Exclusion Criteria:

* Low likelihood of CS/Other explanation for symptoms

  * Inability to consent
  * Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-07-02 (Actual)

PRIMARY OUTCOMES:
Visual interpretation of FDG uptake | 90 minutes
  Images will be evaluated for focal or focal-on-diffuse FDG uptake of the left ventricle or focal RV uptake. The relationship between the location of inflammation and perfusion defects will be characterized ("perfusion metabolism mismatch").
Visual interpretation of FDG uptake | 120 minutes
  Images will be evaluated for focal or focal-on-diffuse FDG uptake of the left ventricle or focal RV uptake. The relationship between the location of inflammation and perfusion defects will be characterized ("perfusion metabolism mismatch").
Severity of myocardial inflammation | 90 minutes
  the maximum standardized uptake value in the heart (cardiac SUV max; g/ml) will be calculated and used to represent the peak level of inflammation.
Severity of myocardial inflammation | 120 minutes
  the maximum standardized uptake value in the heart (cardiac SUV max; g/ml) will be calculated and used to represent the peak level of inflammation.
The extent of inflammation | 90 minutes
  the volume (cm^3) of inflamed myocardium will be calculated using a pre-specified threshold of 2.7 as well as by deriving a unique threshold for each patient by multiplying the background activity x 1.5.
The extent of inflammation | 120 minutes
  the volume (cm^3) of inflamed myocardium will be calculated using a pre-specified threshold of 2.7 as well as by deriving a unique threshold for each patient by multiplying the background activity x 1.5.

SECONDARY OUTCOMES:
Visual interpretation of FDG uptake | 2 weeks after initial scan
  Images will be evaluated for focal or focal-on-diffuse FDG uptake of the left ventricle or focal RV uptake. The relationship between the location of inflammation and perfusion defects will be characterized ("perfusion
Severity of myocardial inflammation | 2 weeks after initial scan
  the maximum standardized uptake value in the heart (cardiac SUV max; g/ml) will be calculated and used to represent the peak level of inflammation.
The extent of inflammation | 2 weeks after initial scan
  the volume (cm^3) of inflamed myocardium will be calculated using a pre-specified threshold of 2.7 as well as by deriving a unique threshold for each patient by multiplying the background activity x 1.5.

CONTACTS AND LOCATIONS:
Overall Officials: Edward J Miller, MD PhD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alvi RM, Young BD, Shahab Z, Pan H, Winkler J, Herzog E, Miller EJ. Repeatability and Optimization of FDG Positron Emission Tomography for Evaluation of Cardiac Sarcoidosis. JACC Cardiovasc Imaging. 2019 Jul;12(7 Pt 1):1284-1287. doi: 10.1016/j.jcmg.2019.01.011. Epub 2019 Mar 4. No abstract available. PMID 30846271